CLINICAL TRIAL: NCT02185872
Title: The Influence of a CrossFit Exercise Program on Glucose Control in Overweight and Obese Individuals
Brief Title: CrossFit Exercise to Improve Glucose Control for Overweight and Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansas State University (Other)
Responsible Party: Principal Investigator, Katie M. Heinrich, Assistant Professor, Kansas State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #6058
Record Dates: First submitted 2014-07-03; First posted 2014-07-10 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Hyperglycemia
Keywords: Exercise; Physical Fitness; Body Composition, Beneficial
MeSH Terms: conditions — Hyperglycemia; Motor Activity; Glucocorticoid Receptor Deficiency | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic and Resistance Training (Active Comparator): Participants completed 24 exercise sessions based on current guidelines. Aerobic exercise (50 min) was performed on machines every session and resistance training (20 min) was performed on machines two sessions per week. Aerobic intensity was prescribed at 40-50% of heart rate reserve (HRR) Weeks 1-4 and 50-60% HRR Weeks 5-8. Resistance training was supervised by an ACE certified personal trainer. One-repetition maximums (1-RM) were assessed Week 1 (i.e., seated bicep curl, military press, seated lat pulldown, seated leg extension, triceps pulldown, bench press, reverse leg curl, seated leg press). For Weeks 2-3 participants completed, 3 sets of 15 reps at 50% 1-RM; Weeks 4-5, 3 sets of 12 reps at 60% 1-RM; Weeks 6-7, 3 sets of 10 reps at 70% 1-RM; Week 8, 3 sets of 8 reps at 75% 1-RM. Three sets of 15 unweighted crunches were completed each day. One minute of rest was taken between each set and each exercise.
  Interventions: Other: Aerobic and Resistance Training
- High-intensity functional training (Experimental): Participants completed a total of 24 sessions that were pre-programmed and led by a certified instructor (CrossFit Level 2), which lasted up to 60 minutes in duration. The first two class periods were structured as an introduction to common movements used in high-intensity functional training (HIFT; e.g., squats, deadlift, press, jerks, barbell, dumbbell, and medicine ball cleans, pullups, kettlebell swings, among others). No scheduled workouts were given on days 1 and 2. Beginning on day 3 each HIFT class consisted of 10-15 minutes of stretching and warmup, 10-20 minutes of instruction and practicing techniques and movements, and 5-30 minutes for the workout of the day, performed at vigorous intensity, relative to each person's ability and fitness level. All weights and movements were individually prescribed and recorded for each participant.
  Interventions: Other: High-Intensity Functional Training

INTERVENTIONS:
Other: High-Intensity Functional Training — Participants were instructed to work as hard as they could while maintaining safe technique and proper form to achieve as many reps or rounds as possible in the prescribed time frame. As HIFT participants became accustomed to specific movements, less time was dedicated to practicing movements and technique.
  Other Names: CrossFit
  Arms: High-intensity functional training
Other: Aerobic and Resistance Training — The protocol was based upon current guidelines of 150 minutes moderate-intensity aerobic activity and 2 days of muscle strengthening per week.
  Arms: Aerobic and Resistance Training

SUMMARY:
The purpose of this study was to examine the differences in glucose control, fitness, and body composition between a standard aerobic and resistance exercise training program and a shorter-duration, high-intensity CrossFit training program in overweight and obese physically inactive adults.

Hypotheses:

1. Both groups would improve glucose control, with the CrossFit group improving significantly more than the aerobic and resistance training group.
2. Both groups would improve fitness, with the CrossFit group improving significantly more than the aerobic and resistance training group.
3. Both groups would demonstrate decreases in body fat percentage and fat mass and increases in lean body mass, with the CrossFit group improving significantly more than the aerobic and resistance training group.

DETAILED DESCRIPTION:
Overweight or obese participants will take part in an 8-week exercise intervention after clearance from a doctor, that is expected to improve glucose control, fitness (Eurofit and peak aerobic capacity), and body composition (body fat percentage, fat mass, and lean body mass). After stratification by age and body mass index, participants will be randomized to either a standard aerobic and resistance training exercise program or a relatively higher intensity, shorter duration CrossFit exercise program.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) of 25 - < 40, physically inactive (i.e., not participating in any structured exercise programs for the past 2 months and not exceeding 30 total minutes of physical activity per week)

Exclusion Criteria:

* current smoker, pregnant, taking blood glucose altering medications, heart disease, type 1 or 2 diabetes mellitus, total cholesterol 200 mg/dL or higher

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-02; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glucose control. | Baseline, Week 10
  Fasting plasma glucose levels were taken after an overnight fast of at least 8 hours. An oral glucose tolerance test was conducted after ingestion of a 75g oral dextrose solution with finger sticks at 30, 45, and 60 minutes from time 0. The following equation was used to calculate glucose area under the curve which was the metric utilized to ascertain changes in glucose control: [(Time 45 - Time 30) * ½ (OGTT 30 + OGTT 45)] + [(Time 60 - Time 45) * ½ (OGTT 60 + OGTT 45)]

SECONDARY OUTCOMES:
Change from baseline in peak aerobic capacity | Baseline, Week 10
  Modified Balke protocol
Change from baseline in sit and reach | Baseline, Week 10
  Eurofit protocol for sit and reach distance using flex tester box
Change from baseline in standing broad jump | Baseline, Week 10
  Eurofit protocol
Change from baseline in vertical jump | Baseline, Week 10
  Eurofit protocol
Change from baseline in pushups | Baseline, Week 10
  Eurofit protocol; completed on feet or knees
Change from baseline in situps | Baseline, Week 10
  Eurofit protocol
Change from baseline in 40 meter dash | Baseline, Week 10
  A handheld stopwatch was used to record time from the command "Go" until the participant crossed the line at 40 meters
Change from baseline in stork balance test | Baseline, Week 10
Change from baseline in body composition | Baseline, Week 12
  Dual X-ray absorptiometry scan was used to assess body fat percentage, lean body mass, and fat mass.

OTHER OUTCOMES:
Time spent completing daily workouts | 24 exercise sessions over 8 weeks
  Time spent to complete each assigned daily workout was individually recorded for each participant

CONTACTS AND LOCATIONS:
Overall Officials: Katie M Heinrich, PhD, Principal Investigator — Kansas State University; Pratik Patel, MS, RD, Study Director — Kansas State University
Locations (1):
- Kansas State University, Manhattan, Kansas, United States

REFERENCES:
- [Result] Heinrich KM, Patel PM, O'Neal JL, Heinrich BS. High-intensity compared to moderate-intensity training for exercise initiation, enjoyment, adherence, and intentions: an intervention study. BMC Public Health. 2014 Aug 3;14:789. doi: 10.1186/1471-2458-14-789. PMID 25086646